Title: Repeated Cannabis Administration on Experimental Pain and Abuse Liability

**NCT:** 04576507

Document date: April 14, 2025

## **Statistical Analysis**

<u>Overview</u>: All data analyses will be based on models using repeated measures analysis of variance (RM-ANOVA) analyzed as a function of cannabis condition (active vs. inactive) and day (Day 1-15), and sets of planned comparisons, calculated with SPSS or SUPERANOVA statistical packages. The planned comparisons are *a priori*, and designed to test the specific hypothesis for each aim. Tests of differences for all comparisons will be based on F-statistics with degrees of freedom corrected, depending on the observed within-subject correlation of the measures, using the method of Geiser and Greenhouse or Huynh and Feldt. Results will be considered statistically significant at p < 0.05, using 2-tailed tests. Distribution of demographic variables (ethnicity, age, sex) will be described in terms of means, standard deviations, proportions, and 95% confidence intervals, where appropriate.